CLINICAL TRIAL: NCT00841685
Title: The Implantation Under Echography of Fiducial Markers in the Intraprostatic Lesion and Prostate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: IBA, Germany (Unknown); Hospimed, Netherland (Unknown); Bard Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2008/109
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): Goldlock
  Interventions: Device: Goldlock
- 2 (Active Comparator): Visicoil smallest size
  Interventions: Device: Visicoil smallest size
- 3 (Active Comparator): Visicoil larger size
  Interventions: Device: Visicoil larger size
- 4 (Active Comparator): Bard goldmarker smallest size
  Interventions: Device: Bard goldmarker smallest size
- 5 (Active Comparator): Bard goldmarker larger size
  Interventions: Device: Bard goldmarker larger size

INTERVENTIONS:
Device: Goldlock — Insertion of Goldlock marker
  Arms: 1
Device: Visicoil smallest size — Insertion of Visicoil, smallest size, marker
  Arms: 2
Device: Visicoil larger size — Insertion of Visicoil, larger size, marker
  Arms: 3
Device: Bard goldmarker smallest size — Insertion of Bard goldmarker, smallest size
  Arms: 4
Device: Bard goldmarker larger size — Insertion of Bard goldmarker, larger size
  Arms: 5

SUMMARY:
Implantation of fiducial markers in the prostate and daily check of the positioning during radiotherapy based on the implanted fiducial markers

ELIGIBILITY:
Inclusion Criteria:

* histological proven adenocarcinoma of the prostate
* T1-T4 tumors
* Radiotherapy as primary therapy +/- androgen deprivation
* Presence of an intraprostatic lesion (IPL) on MRI/MRS
* Presence of an intraprostatic lesion (IPL) on ultrasound
* WHO 0-2

Exclusion Criteria:

* Other primary tumor, except non-melanoma skin cancer
* No written informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2012-05-01 (Actual); Study Completion 2012-05-01 (Actual)

PRIMARY OUTCOMES:
Acute toxicity after implantation of the fiducial gold markers | 1 week after implantation

SECONDARY OUTCOMES:
Feasibility of insertion 1 fiducial gold marker in the intraprostatic lesion combined with extra gold markers in the rest of the prostate upto 3 goldmarkers in total | 1 week after implantation
Visualization of the implanted gold markers by ultrasound | After implantation

CONTACTS AND LOCATIONS:
Overall Officials: Gert De Meerleer, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be